CLINICAL TRIAL: NCT01297673
Title: Vesico-ureteral Reflux in a Contemporary Series of Spinal Cord Injury Patients With Neurogenic Lower Urinary Tract Dysfunction
Brief Title: Reflux in Spinal Cord Injury Patients With Neurogenic Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Kessler, PD Dr. med., Balgrist University Hospital
Other Study IDs: EK 2010-0207/02
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Vesico-ureteral Reflux; Spinal Cord Injury
Keywords: vesico-ureteral reflux; neurogenic bladder dysfunction; spinal cord injury
MeSH Terms: conditions — Vesico-Ureteral Reflux; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal cord injury: Patients with neurogenic lower urinary tract dysfunction due to spinal cord injury with regular urodynamic examination
  Interventions: Procedure: video-urodynamic examination

INTERVENTIONS:
Procedure: video-urodynamic examination — Assessment of bladder function during video urodynamic determine of incidence degree and localization of vesico ureteral reflux based on the result of video urodynamics

SUMMARY:
The purpose of this study is to investigate the incidence of reflux in patients with spinal cord injury in relation to the lesion level, duration of injury and bladder management

DETAILED DESCRIPTION:
Vesico-ureteral reflux was the main cause for renal failure and reduced life expectancy in patients with neurogenic bladder dysfunction due to spinal cord injury. Neurogenic detrusor overactivity leads to high intravesical pressure and may induce reflux. Decreasing intravesical pressure and increasing bladder capacity is necessary to prevent reflux and secondary renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* Neurogenic lower urinary tract dysfunction
* Written informed consent

Exclusion Criteria:

* Lower urinary tract dysfunction due to other causes than spinal cord injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages Eligibility: minimum 18 years Genders Eligibility: female and male
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence and degree of vesico ureter renal reflux | average: yearly scheduled control
  video urodynamic, ultrasound examination

SECONDARY OUTCOMES:
pdet (cmH2O) | average: yearly scheduled control
  urodynamic parameter, detrusor pressure
Medication | average: yearly scheduled examination
  name of drugs and applied dosis
possible complications | average: yearly scheduled examination
  urinary tract infection, pyelonephritis, renal dysfunction
maximum cystometric capacity | average: yearly scheduled control
  the volume at which a patient, with normal sensation, fells he/she can no longer delay micturition
compliance mL/cmH2O | average: yearly scheduled control
  Compliance is the change in volume divided by change in detrusor pressure expressed as mL/cmH2O.
bladder management | average: yearly scheduled control
  most common: intermittent catheterisation, indwelling catheter, external condom urinal for male patients

CONTACTS AND LOCATIONS:
Locations (1):
- Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland